CLINICAL TRIAL: NCT04409067
Title: The Use of Electromyography in the Assessment of Masticatory Muscle Activity in Patients With Pain-related Temporomandibular Disorders
Brief Title: Masticatory Muscle Activity in Patients With Pain-related Temporomandibular Disorders
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Liliana Szyszka-Sommerfeld, DDS, PhD, Pomeranian Medical University Szczecin
Other Study IDs: 0012/08/15
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: TMD
Keywords: masticatory muscles; surface electromyography; muscle activity
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TMD-pain group: The TMD-pain group consisted of 30 children aged between 7.1 and 12.3 with a pain-related TMD diagnosis. All the patients in the TMD-pain group had myogenous or arthrogenous TMD according to the RDC/TMD protocol.
  Interventions: Diagnostic Test: electromyography
- pain-free TMD group: The pain-free TMD group consisted of 30 children between 7.3 and 12.6 years of age. To be included in the pain-free TMD group the participants had to meet Axis I of the RDC/TMD criteria for a pain-free diagnosis.
  Interventions: Diagnostic Test: electromyography
- non-TMD group: The non-TMD group comprised 30 children aged between 7.2 and 12.5 without any recognised TMD based on RDC/TMD, Axis I.
  Interventions: Diagnostic Test: electromyography

INTERVENTIONS:
Diagnostic Test: electromyography — Surface electromyography (sEMG) was used as an additional non-invasive tool for assessing patients with TMD.The electromyographical (EMG) potentials of the temporalis and masseter muscles were measured with a DAB-Bluetooth Instrument (Zebris Medical GmbH, Germany) at rest and during maximum voluntary clenching (MVC).

SUMMARY:
The aim of this study was to evaluate masticatory muscle electrical activity in patients with pain-related and pain-free temporomandibular disorders (TMD) as well as in subjects with no TMD. Ninety children with mixed dentition were recruited to the study. Of this total, 30 subjects were diagnosed with pain-related TMD, 30 with pain-free TMD, and 30 without TMD. We used Axis I of the Research Diagnostic Criteria for TMD (RDC/TMD) to assess the presence of TMD in the examined children. The electromyographical (EMG) potentials of the temporalis and masseter muscles were measured with a DAB-Bluetooth Instrument (Zebris Medical GmbH, Germany) at rest and during maximum voluntary clenching (MVC).

ELIGIBILITY:
Inclusion Criteria:

* mixed dentition (the subjects should be aged between 7 and 12 years)
* consent to participate voluntarily in the study

Exclusion Criteria:

* subjects who had undergone orthodontic or masticatory motor system dysfunction treatment, had systemic or rheumatologic diseases, a history of mouth breathing, surgery, traumas or malformations in the head and neck region

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The subjects were selected from patients who had been referred to the Orthodontic Clinic in Szczecin, Poland for orthodontic treatment.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Electromyographic analysis of the masticatory muscles in patients with pain-related temporomandibular disorders | For a single subject the whole EMG examination was taken 40 minutes.
  A DAB-Bluetooth Instrument (Zebris Medical GmbH, Germany) was used to take electromyographical (EMG) recordings of the temporalis and masseter muscles at rest and during maximum voluntary contraction (MVC).Disposable, self-adhesive Ag/AgCl bipolar surface electrodes were placed at a fixed inter-electrode distance of 20 mm on the anterior temporal muscles and on the superficial masseter muscles parallel to the muscular fibres. The EMG signals were amplified, digitized and digitally filtered. The EMG results were analysed using the Student t-test, analysis of variance (ANOVA) and a Student-Newman-Keuls post-hoc test.

CONTACTS AND LOCATIONS:
Locations (1):
- Pomeranian Medical University, Department of Orthodontics, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided